CLINICAL TRIAL: NCT05499598
Title: Clinical and Radiographic Evaluation of Modified Minimally Invasive Surgical Technique and Platelet Rich Fibrin With or Without Vitamin Pool A and C for Management of Periodontal Intrabony Defects: A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Modified Minimally Invasive Surgical Technique and Platelet Rich Fibrin With or Without Vitamin Pool A and C for Management of Periodontal Intrabony Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dalia Sanaa Abdel Ghaffar, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PERAUG2022
Record Dates: First submitted 2022-08-11; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Intrabony Periodontal Defect
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified minimally invasive surgical technique with PRF and vitamins A and C (Experimental): Surgical technique (M-MIST) with the same procedures will be performed. Approximately 10 mm of fresh blood will be drawn by venipuncture of the antecubital vein and collected into a blood collection tube without anticoagulant. Ascorbic Acid will be added to the fresh blood to achieve a concentration of 250 μg/ml, Retinol will also be added to achieve a concentration of 20 μmol/L. The resultant PRF clot will be placed into the intra-osseous defect.
  Interventions: Procedure: Experimental: Modified minimally invasive surgical technique with PRF and vitamins A and C
- Modified minimally invasive surgical technique with PRF (Active Comparator): Surgical technique (M-MIST) with the same procedures will be performed. Approximately 10 mm of whole blood is drawn by venipuncture of the antecubital vein and is collected into two blood collection tubes without anticoagulant for PRF preparation.The resultant PRF clot will be placed into the intra-osseous defect
  Interventions: Procedure: Modified minimally invasive surgical technique with PRF

INTERVENTIONS:
Procedure: Experimental: Modified minimally invasive surgical technique with PRF and vitamins A and C — Surgical technique (M-MIST) with the same procedures will be performed. Approximately 10 mm of fresh blood will be drawn by venipuncture of the antecubital vein and collected into a blood collection tube without anticoagulant. Ascorbic Acid will be added to the fresh blood to achieve a concentration of 250 μg/ml, Retinol will also be added to achieve a concentration of 20 μmol/L. The resultant PRF clot will be placed into the intra-osseous defect.
  Arms: Modified minimally invasive surgical technique with PRF and vitamins A and C
Procedure: Modified minimally invasive surgical technique with PRF — Surgical technique (M-MIST) with the same procedures will be performed. Approximately 10 mm of fresh blood will be drawn by venipuncture of the antecubital vein and collected into a blood collection tube without anticoagulant. The resultant PRF clot will be placed into the intra-osseous defect.
  Arms: Modified minimally invasive surgical technique with PRF

SUMMARY:
This study aims to assess clinical and radiographic outcomes after the use of vitamins A and C with PRF versus PRF alone in the treatment of periodontal intrabony defect.

DETAILED DESCRIPTION:
Sites with deep intrabony defects were considered to be at a higher risk of disease progression if patients did not receive any systematic periodontal therapy. Treatment of intrabony defects is an important therapeutic goal of periodontal therapy. The optimal outcome of treatment in intrabony defects is considered to be the absence of bleeding on probing, the presence of shallow pockets associated with periodontal regeneration and limited soft tissue recession.The minimally invasive surgical technique is designed to mobilize just the defect-associated papilla and to reduce flap extension as much as possible. The modified minimally invasive surgical technique has been proposed to further reduce invasiveness and patient side effects by limiting the incision line to the buccal side. This technique fulfilled the maintenance of the interdental papillary height by minimizing its tendency to collapse, increased the likelihood of primary wound closure and reduced the chances of gingival recession.

Platelet-rich fibrin is a powerful healing biomaterial with inherent regenerative capacity and can be used in the treatment of periodontal intrabony defects.

Vitamin C is found to be able to induce osteogenic differentiation and maturation of progenitor cells of PDL without using osteogenic filling material. Also, Vitamin A has a unique property of de-differentiating adult cells into pluripotent cells.

Since combination therapies have been shown to be effective in the regeneration of periodontal defects, this study will evaluate the synergetic effect of vitamins A and C on the periodontal regeneration, together with the most widely used regenerative biomaterial; Platelet-rich fibrin, as an attempt for finding the gold standard in the treatment of intra-bony defects.

ELIGIBILITY:
Inclusion Criteria:

* Patient-related criteria:

  * Patient consulting in the outpatient clinic with periodontitis stage III
  * Able to tolerate surgical periodontal procedures.
  * Patient ready to perform oral hygiene instructions.
  * Compliance with the maintenance program.
  * Provide informed consent.
  * Accepts the 6 months follow-up period.

Teeth related criteria:

* Mature permanent tooth.
* Tooth with two or three-walled intra-bony defect, with CAL ≥ 5mm and intra osseous defect ≥ 3mm.

Exclusion Criteria:

* Patient-related criteria:

  * Medically compromised patients.
  * Pregnant or nursing women.
  * Uncooperative patients.
  * Smokers.

Teeth related criteria:

* Teeth with one wall intra-bony defect.
* Teeth with supra-bony defects.
* Teeth with grade III mobility.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Radiographic linear defect depth (mm) | 9 months
  Digital Radiographs using ImageJ software, Measured as the depth of intra-osseous defect from the alveolar crest to the defect.

SECONDARY OUTCOMES:
Probing depth (mm) | 9 months
  Measured from the gingival margin to the bottom of the gingival sulcus
Clinical Attachment Level (mm) | 9 months
  Measured from the CEJ to the bottom of the gingival sulcus
Gingival Recession Depth (mm) | 9 months
  Measured from the CEJ to the most apical extension of the gingival margin

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heitz-Mayfield LJ, Lang NP. Surgical and nonsurgical periodontal therapy. Learned and unlearned concepts. Periodontol 2000. 2013 Jun;62(1):218-31. doi: 10.1111/prd.12008. PMID 23574468
- [Background] Elbehwashy MT, Hosny MM, Elfana A, Nawar A, Fawzy El-Sayed K. Clinical and radiographic effects of ascorbic acid-augmented platelet-rich fibrin versus platelet-rich fibrin alone in intra-osseous defects of stage-III periodontitis patients: a randomized controlled clinical trial. Clin Oral Investig. 2021 Nov;25(11):6309-6319. doi: 10.1007/s00784-021-03929-1. Epub 2021 Apr 12. PMID 33842996
- [Background] Fawzy El-Sayed KM, Hein D, Dorfer CE. Retinol/inflammation affect stemness and differentiation potential of gingival stem/progenitor cells via Wnt/beta-catenin. J Periodontal Res. 2019 Aug;54(4):413-423. doi: 10.1111/jre.12643. Epub 2019 Mar 4. PMID 30830694
- [Background] Dohan DM, Choukroun J, Diss A, Dohan SL, Dohan AJ, Mouhyi J, Gogly B. Platelet-rich fibrin (PRF): a second-generation platelet concentrate. Part I: technological concepts and evolution. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Mar;101(3):e37-44. doi: 10.1016/j.tripleo.2005.07.008. Epub 2006 Jan 19. PMID 16504849